CLINICAL TRIAL: NCT07161726
Title: Cocoa to Maximize Exercise Training in Older Adults - The COMET Trial
Acronym: COMET
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Robert T Mankowski, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-300015048
Record Dates: First submitted 2025-09-02; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Mobility Disability
Keywords: Cocoa; Exercise; Mobility; Older adults
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (-)-Epicatechin combined with exercise (Active Comparator): 12 weeks of daily cocoa (2 capsules/d containing 450 mg cocoa flavanols/d, including 80 mg of (-)-epicatechin) combined with aerobic (30min of moderate-intensity walking) and resistance (25 min of whole-body workout) exercise training 3 times a week
  Interventions: Combination Product: (-)-Epicatechin-rich cocoa supplementation combined with exercise training
- Placebo combined with exercise (Placebo Comparator): 12 weeks of placebo (alike-looking cellulose-based capsules) combined with aerobic (30min of moderate-intensity walking) and resistance (25 min of whole-body workout) exercise training 3 times a week
  Interventions: Combination Product: Placebo combined with exercise training

INTERVENTIONS:
Combination Product: (-)-Epicatechin-rich cocoa supplementation combined with exercise training — 12 weeks of daily cocoa (2 capsules/d containing 450 mg cocoa flavanols/d, including 80 mg of (-)-epicatechin) combined with aerobic (30min of moderate-intensity walking) and resistance (30 min of whole-body workout) exercise training 3 times a week
  Arms: (-)-Epicatechin combined with exercise
Combination Product: Placebo combined with exercise training — 12 weeks of placebo (alike-looking cellulose-based capsules) combined with aerobic (30min of moderate-intensity walking) and resistance (30 min of whole-body workout) exercise training 3 times a week
  Arms: Placebo combined with exercise

SUMMARY:
The purpose of the study is to see if regular exercise when combined with a cocoa supplement will improve physical performance and muscle strength compared to regular exercise alone.

DETAILED DESCRIPTION:
Diminished mitochondrial function, excessive production of reactive oxygen species (ROS) and mitochondrial DNA (mtDNA) damage are key contributors to age-related physical capacity and muscle strength decline. Adaptation to aerobic and strength exercise training is currently one of the most effective ways to preserve physical performance and muscle strength in older adults. Aerobic and resistance exercise training improves mitochondrial function and stabilizes production of ROS, which contribute to aerobic capacity as well as strength improvements. However, obtaining optimal effects of exercise training may be limited by heterogeneity in the responsiveness due to biological barriers in skeletal muscle energy production, regardless of the adherence. Therefore, there is an unmet need for combining non-pharmacologic therapies with exercise training to "unlock" its full energetic potential to more effectively improve physical performance and muscle strength in older adults at risk of mobility disability. (-)-Epicatechin, a flavanol and a major ingredient present in cocoa, improved survival, muscle mitochondrial function and reduced excess ROS in mice. Supplementation with (-)-epicatechin-rich cocoa improved walking performance and muscle strength in older adults. Combination of (-)-epicatechin with exercise further improved mitochondrial function and reduced muscle fatigue in mice. We hypothesize that the combination of (-)-epicatechin-rich cocoa with structured aerobic and resistance exercise training will be more effective than exercise alone in improving physical performance and muscle strength by improved mitochondrial function and reduced ROS production in moderately functioning older adults. Our proposed pilot trial will test a 3-month exercise training intervention to collect preliminary data on walking performance, muscle strength and muscle size in 36 moderately functioning (slow walking speed <1m/s) older adults (>55 years old) without major comorbidities. The participants will be randomized to 12-week of daily (-)-epicatechin-rich cocoa (2 capsules/d containing 450 mg cocoa flavanols/day, including 80 mg of (-)-epicatechin) combined with aerobic (30min of moderate-intensity walking) and resistance (25 min of whole-body workout) exercise training 3 times a week (Epi+Ex, n=18) or the same exercise training regimen combined with cellulose-based blind (PL+Ex, n=18). Our primary outcome is walking distance measured by the 6-minute walk test. The lower-limb muscle strength and size measured by the Biodex test will be our secondary outcome. We will explore the potential mechanism of the hypothesized effect of Epi+Ex on walking performance and muscle strength by measuring mitochondrial biogenesis, mitochondrial DNA damage, ROS production and antioxidant enzyme activity in the vastus lateralis biopsies at baseline and 12-week follow-up. The objective of this exploratory/developmental proposal is to gather preliminary data on the efficacy and explore the mechanism of the Epi-Ex intervention to support the future Phase II clinical trial testing (-)-epicatechin-rich cocoa flavanols for exercise training optimization in older adults.

ELIGIBILITY:
Inclusion Criteria:

* Age 55 years and older
* Slow walking speed of < 1m/s
* Willingness to be randomized to either treatment group
* Willingness to participate in all study procedures (muscle biopsy will be optional)

Exclusion Criteria:

* Failure to provide informed consent;
* Regular consumption of flavanol and/or cocoa supplements
* Current involvement in supervised rehabilitation/exercise training program
* Absolute contraindication(s) to exercise training according to American College of Sports Medicine guidelines [17]
* Daytime average of systolic blood pressure ≥ 180/100mm Hg.
* Refusal to stop blood thinners such as baby aspirin dose.
* Peripheral vascular disease; peripheral neuropathy; retinopathy
* Severe cardiac disease, including NYHA Class III or IV congestive heart failure, clinically significant aortic stenosis, history of cardiac arrest, use of a cardiac defibrillator, or uncontrolled angina;
* Myocardial infarction or stroke within past year
* Significant cognitive impairment, including known dementia diagnosis or a Mini-Mental State Examination exam score < 24
* Progressive, degenerative neurologic disease, e.g., Parkinson's Disease, multiple sclerosis;
* Severe rheumatologic or orthopedic diseases, e.g., awaiting joint replacement, active inflammatory disease;
* Severe pulmonary disease, requiring either steroid pills or injections or the use of supplemental oxygen;
* Hip fracture, hip or knee replacement, or spinal surgery within past 4 months;
* Other significant co-morbid conditions that would impair ability to participate in the exercise-based intervention
* Simultaneous participation in another interventional trial

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
6-min walk test | At the baseline, 6-week, and 12-week follow-up visits.
  We will assess exercise capacity of participants using the 6-min walk test, a safe and reliable test of aerobic endurance in older persons. This test has strong reproducibility, with intra-subject coefficients of variation averaging < 10%, and has a modest correlation with peak VO2peak. Participants will be asked to walk as far and fast as possible for 6-min on a 60 m distance making u-turns at 60m and start line cones.

SECONDARY OUTCOMES:
Biodex test | At the baseline, 6-week, and 12-week follow-up visits.
  Maximal strength (peak torque) of the knee flexors and extensors of the dominant limb will be assessed by a dynamometer (Biodex Medical Systems, New York, NY) as published previously. Based on our long-standing experience in performing muscle strength Biodex tests, these tests are reliable in moderately functioning older adults and are well-tolerated.

CONTACTS AND LOCATIONS:
Overall Officials: Robert T Mankowski, PhD, Principal Investigator — University of Alabama at Birmingham

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data may not be shared due to privacy concerns, the risk of re-identification in a small cohort, and the absence of participant consent for external data sharing.